CLINICAL TRIAL: NCT06674447
Title: Awareness Among Physical Therapists Of Baluchistan Regarding Effectiveness Of Sensory Integration Therapy On Cerebral Palsy Population
Brief Title: Awareness Among PT Regarding Sensory Integration Therapy on CP Population
Status: Recruiting | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCH&AHS/24/ayesha waqar
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Sensory Integration Disorder (Disorder)
Keywords: Cerebral Palsy; sensory integration disorder
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is to interrogate the awareness level of physiotherapists that are working in the region of Baluchistan, to access weather know about sensory integration therapy or they use it for the patients of cerebral palsy in their treatment plan or not.

DETAILED DESCRIPTION:
The study title is ''AWARENESS AMONG PHYSICAL THERAPISTS OF BALUCHISTAN REGARDING EFFECTIVENESS OF SENSORY INTEGRATION THERAPY ON CEREBRAL PALSY POPULATION.' it is a cross-sectional study that will be conducted in the province of Baluchistan, Pakistan. The data will be conducted by 200 physical therapists on a self designed tool, that will allows us to know about the awareness among the physical therapist of this particular region to know if they are using sensory integration therapy in the treatment plan of the children suffering from cerebral palsy to know weather the sensory issues are being addressed over there by this therapy or not. Another purpose of this study is to make the therapists aware about sensory integration therapy and its efficacy in treating sensory processing and sensory integration issues present in the children that are suffering from cerebral palsy. The data will be collected by the physical therapists that are currently working in various hospitals of Baluchistan located in different regions of the province.

ELIGIBILITY:
Inclusion Criteria: Physical therapists working in province of Baluchistan, specifically.

Exclusion Criteria: Physical therapists working in areas other than Baluchistan.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The Physical therapists of Baluchistan, that are exclusively practising in various areas of Baluchistan.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Survey tool awareness of PT,s about Sensory Integration therapy | 20 minutes
  survey was conducted through adapted questionnaire among the physiotherapist of Baluchistan

CONTACTS AND LOCATIONS:
Overall Officials: AYESHA WAQAR, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hume K, Steinbrenner JR, Odom SL, Morin KL, Nowell SW, Tomaszewski B, Szendrey S, McIntyre NS, Yucesoy-Ozkan S, Savage MN. Evidence-Based Practices for Children, Youth, and Young Adults with Autism: Third Generation Review. J Autism Dev Disord. 2021 Nov;51(11):4013-4032. doi: 10.1007/s10803-020-04844-2. Epub 2021 Jan 15. PMID 33449225